CLINICAL TRIAL: NCT02264899
Title: MEMENTO-VAScular COmponents of Dementia
Acronym: VASCOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2012/32
Record Dates: First submitted 2014-10-01; First posted 2014-10-15 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Alzheimer's Disease (AD); Alzheimer's Disease (AD) Related Disorders
Keywords: Alzheimer's disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alzheimer's disease and related disorders (Experimental)
  Interventions: Other: in Memento-VASCOD

INTERVENTIONS:
Other: in Memento-VASCOD — * Pulse wave velocity assessment
  * Cerebral MRI including Arterial Spin Labeling (ASL) and Magnetic Resonance Angiography (MRA) sequences
  * Ophthalmological exams: Spectral Domain-Optical Coherence Tomography (SD-OCT), colour photographs of the retina, visual acuity and axial lenght measurement
  * Neuropsychological testing and behaviorial and mood scales
  * Urinary albumin excretion measurement

SUMMARY:
A Multicenter national longitudinal cohort study including at least 800 individuals recruited from French Research Memory Centers and followed up over 36 months and included in Memento.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a neurodegenerative disorder thought to be caused by the accumulation of the peptide amyloid beta and the hyperphosphorylated tau protein in the brain. There are increasing arguments in favor of an important role of vascular damages in the development and progression of AD.

The time course of these vascular alterations and how they relate to dementia and AD pathology remain unclear, as no protocol that allows the development of the diverse vascular pathology to be scored, and hence to be tracked with ageing, has so far been developed and widely validated. The aims of this project are to investigate, in a large clinical sample of patients presenting either isolated cognitive complaints or light to mild cognitive deficits, how vascular risk factors and vascular alterations (assessed at macro and micro levels) relate to cerebrovascular disease and cognitive decline.

The primary objective of this ancillary study is to investigate the prospective association between vascular risk factors, inflammation markers and vascular damages on cognitive decline and neurodegeneration progression over up to 4 years of follow-up in a sample of individuals presenting with a spectrum of cognitive profiles ranging from isolated cognitive complaints to cognitive deficits without dementia.

The secondary objectives are the following

* To investigate the role of vascular risk factors (diabetes, hypertension, hypercholesterolemia) and vascular damages on progression to clinical dementia over up to 4-year follow-up.
* To study whether the interaction between changes in markers of macrovascular and microvascular structures on cognitive deficits progression.
* To study the association between in BP, hypertension, antihypertensive treatments and vascular damages, progression of cerebrovascular disease seen at MRI and cognitive decline and dementia risk
* To assess the temporality of vascular damages burden on neurodegeneration
* To assess the association between retinal vasculature defect and brain neurovascular damages
* To study the link between vascular damages and AD pathology (Cerebro-Spinal Fluid (CSF) and Positron emission tomography (TEP) amyloid imaging) biomarkers in the subsample of participants having all measures available
* To investigate how inflammatory markers mediate the association between vascular damages and neurodegeneration
* To assess whether vascular factors and neurodegenerative factors act independently or synergistically on the course of cognitive decline
* To assess simultaneously the impact of vascular damages on end organs (brain, eye, and kidney)
* To study the correlation between cerebral blood flow, measured by Arterial spin-Labeled (ASL) MRI and cognitive decline
* To study whether genetic polymorphisms revealed from genome-wide association studies (GWAS) of AD of vascular factors could modulate the association between vascular damages and cognitive decline

ELIGIBILITY:
Inclusion Criteria:

* Participants to MEMENTO-Vascod should be included in MEMENTO.
* To have signed a specific MEMENTO-Vascod informed consent form, prior to any Vascod ancillary study related procedures
* To be aged 50 years old and above
* To have a Clinical Dementia Rating scale <0.5 and to be not demented;

Exclusion Criteria:

* Are under guardianship
* Live in skilled nursing facility
* Are Pregnant or breast feeding women
* Meet brain MRI exclusion criteria (Same criteria as in Memento main protocol)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Change in cognitive performances over | 36 months from baseline

SECONDARY OUTCOMES:
Progression to clinical dementia of Alzheimer's type according to standardized criteria | 36 months from baseline
  standardized criteria : Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and National Institute of Neurological and Communicative Disorders and Stroke Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) classifications
Change in CSF and blood amyloid biomarkers of AD | 24 months from baseline
Change in brain atrophy and hippocampal volumes | 24 months from baseline
Progression of small vessels disease markers (white matter lesions, lacunar infarcts, microbleeds) | 24 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve CHENE, Prof, Principal Investigator — CIC-EC1401 - ISPED - CHU de Bodeaux; Geneviève CHENE, Prof, Study Chair — CIC-EC1401 - ISPED - CHU de Bordeaux; Carole DUFOUIL, Director, Study Director — CIC-EC1401 - ISPED - CHU de Bordeaux
Locations (10):
- France (10):
  - CHU d'Amiens, Amiens
  - CHU de Bordeaux - Pellegrin, Bordeaux
  - CHU de Dijon, Dijon
  - CHU de Lille, Lille
  - Hospices civils de Lyon, Lyon
  - AP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - AP-HP - Hôpital BROCA, Paris
  - AP-HP - Hôpital LARIBOISIERE, Paris
  - CHU de Strasbourg, Strasbourg